CLINICAL TRIAL: NCT00246740
Title: Protection of the Heart With Doxycycline During Coronary Artery Bypass Grafting: A Pilot Study
Brief Title: Protection of the Heart With Doxycycline During Coronary Artery Bypass Grafting
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Barry Finegan, Professor, University of Alberta
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Protect Study Protocol
Record Dates: First submitted 2005-10-28; First posted 2005-10-31 (Estimated); Results first posted 2017-12-15 (Actual); Last update posted 2017-12-15 (Actual); Status verified 2017-05

CONDITIONS: Coronary Artery Bypass Grafting; Cardiopulmonary Bypass; Reperfusion Injury
Keywords: Doxycycline; coronary artery bypass grafting
MeSH Terms: conditions — Reperfusion Injury | interventions — Doxycycline

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo oral tablet (Placebo Comparator): Patients received oral administration of matching placebo pills, twice a day at least 2 days prior to surgery, on the day of surgery, and for the first 3 postoperative days (via a nasogastric tube or orally when patients tolerated it).
  Interventions: Drug: Placebo Oral Tablet
- Periostat (Experimental): Patients received oral administration of 20 mg of doxycycline, twice a day at least 2 days prior to surgery, on the day of surgery, and for the first 3 postoperative days (via a nasogastric tube or orally when patients tolerated it).
  Interventions: Drug: Periostat

INTERVENTIONS:
Drug: Periostat — In addition to standard care, patients received oral administration of 20 mg of doxycycline twice a day at least 2 days prior to surgery, on the day of surgery, and on postoperative days 1, 2, and 3.
  Other Names: Doxycycline
  Arms: Periostat
Drug: Placebo Oral Tablet — In addition to standard care, patients received oral administration of placebo twice a day at least 2 days prior to surgery, on the day of surgery, and on postoperative days 1, 2, and 3.
  Other Names: Placebo
  Arms: Placebo oral tablet

SUMMARY:
The purpose of this study is to determine whether doxycycline (Periostat) at a sub-antimicrobial dose will decrease reperfusion injury after coronary artery bypass grafting (CABG) surgery with cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
This proposal is for a randomized, placebo-controlled, double-blinded study of the use of doxycycline in patients requiring CABG surgery. Patients will be randomized 1:1 to receive either doxycycline or placebo.

This study will be conducted in a blinded manner. The pharmacy will randomize patients and will have the randomization code. The code will only be broken in the case of an emergency and the event will be fully documented.

In addition to standard care, patients will receive oral administration of 20 mg of doxycycline or placebo twice a day at least 2 days prior to surgery, on the day of surgery, and on postoperative days 1, 2, and 3.

Myocardial atrial biopsies will be taken at 2 time points during the CABG procedure: during cannulation of the right atrium and 10 minutes after cross-clamp release. Tissue will be analyzed for MMP-2 and -9 activity and TnI and MLC-1 levels.

A Swan-Ganz-Catheter will be placed in the pulmonary artery over 24 hours to measure hemodynamics (LVSWI).

A coronary sinus catheter will be placed under echocardiographic guidance prior to initiation of CPB (will be removed 20 minutes after cross-clamp release).

Patients will have an additional ECG on post-operative days 1 and 3.

Additional blood will be drawn to determine doxycycline plasma levels, MMP-2 and -9 activity, total gelatinolytic activity, and levels of troponin I and T products at the following time points: pre-induction, prior to initiation of CPB, 10 and 20 minutes following the release of the aortic cross clamp (arterial and venous) and 3, 6, 24 and 72 hours post aortic cross clamp removal (venous). Each of the above samples will require 6 mL of blood for a study total of 72 mL. At the time of each blood draw we will measure and record the hematocrit value.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent
* Aged 18 through 80 years, inclusive
* Scheduled for primary CABG surgery with CPB

Exclusion Criteria:

* Females of childbearing potential
* Emergency CABG
* Previous sternotomy
* Planned simultaneous surgery (i.e. valve repair or carotid endarterectomy)
* Myocardial infarction within 48 hours
* Pre-operative atrial fibrillation
* Pre-operative ventricular pacing or left bundle branch block (LBBB)
* Known hypersensitivity to tetracycline class antibiotics
* Renal failure requiring dialysis

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2005-10; Primary Completion 2008-05 (Actual); Study Completion 2009-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Barry A Finegan, FFARCS FRCPC, Principal Investigator — Department of Anesthesiology and Pain Medicine, University of Alberta Hospital
Locations (1):
- University of Alberta Hospital, Edmonton, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Schulze CJ, Castro MM, Kandasamy AD, Cena J, Bryden C, Wang SH, Koshal A, Tsuyuki RT, Finegan BA, Schulz R. Doxycycline reduces cardiac matrix metalloproteinase-2 activity but does not ameliorate myocardial dysfunction during reperfusion in coronary artery bypass patients undergoing cardiopulmonary bypass. Crit Care Med. 2013 Nov;41(11):2512-20. doi: 10.1097/CCM.0b013e318292373c. PMID 23928836
- See also: DOI of published results paper — https://dx.doi.org/10.1097/CCM.0b013e318292373c

RESULTS

PARTICIPANT FLOW:
Period: Initial Enrollment
Arm/Group | Placebo Oral Tablet | Periostat
Started | 28 | 28
Completed | 22 | 20
Not Completed | 6 | 8
Not completed — Death | 1 | 0
Not completed — Additional surgery scheduled | 0 | 2
Not completed — Surgery schedule change | 4 | 4
Not completed — Other | 1 | 2
Period: Experimental Phase
Arm/Group | Placebo Oral Tablet | Periostat
Started | 22 | 20
Completed | 22 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Oral Tablet | Periostat | Total
Number analyzed (Participants) | 22 | 20 | 42
Age, Continuous [Mean (Standard Deviation); unit: years] | 64.6 (1.5) | 63.1 (2) | 63.9 (1.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 3 | 9
  Male | 16 | 17 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 22 | 20 | 42

OUTCOME MEASURES:

1. Primary Outcome: Left Ventricular Stroke Work Index (LVSWI)
Description: Measure of global left ventricular function. The formula used for calculation is: LVSWI= SI x MAP x 0.0144 LVSWI = Left Ventricular Stroke Work Index (g*m/m2) SI = Stroke Index (mL/beat/m2) MAP = Mean Arterial Pressure (mmHg) 0.0144 is a conversion term to equalize units.
Time Frame: Before surgery up to 24h of reperfusion
Measure: Mean (Standard Error); unit: g*m/m2
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
g*m/m2
  Before surgery | 42 (2.6) | 43 (2.5)
  Post surgery | 29 (1.7) | 28 (1.7)
  1h reperfusion | 30 (1.8) | 29 (1.9)
  3h reperfusion | 31 (1.9) | 29 (2)
  6h reperfusion | 28 (1.4) | 25 (1.4)
  12h reperfusion | 30 (1.6) | 30 (1.7)
  24h reperfusion | 32 (1.8) | 33 (1.9)

2. Secondary Outcome: Cardiac Matrix Metalloproteinase-9 Activity in Right Atrial Biopsies at 10 Minutes Reperfusion
Description: Biochemical activity of MMP-9 activity in right atrial biopsies, measured at 10 minutes of reperfusion after surgery. To determine MMP-9 activity, 20 μg of total protein from both myocardial extracts and plasma were analyzed by gelatin zymography. For detailed methodology consult Cheung PY, Sawicki G, Wozniak M, et al: Matrix metalloproteinase-2 contributes to ischemia-reperfusion injury in the heart. Circulation 2000; 101:1833-1839
Time Frame: Before surgery and 10 minutes reperfusion after surgery
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
Arbitrary units
  Before surgery | .75 (.25) | 1.56 (.26)
  10 min reperfusion | .44 (.28) | 1.63 (.29)

3. Secondary Outcome: Cardiac Matrix Metalloproteinase-2 Activity in Right Atrial Biopsies at 10 Minutes Reperfusion
Description: Biochemical activity of MMP-2 activity in right atrial biopsies, measured at 10 minutes of reperfusion after surgery.
Time Frame: Before surgery and 10 minutes reperfusion after surgery
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
Arbitrary units
  Before surgery | .36 (.04) | .24 (.04)
  10 min reperfusion | .42 (.04) | .25 (.04)

4. Secondary Outcome: Venous Plasma Cardiac Matrix Metalloproteinase-9 Activity Before and After Reperfusion
Description: Biochemical activity of MMP-9 activity in venous plasma, measured before surgery and up to 72h of reperfusion after surgery.
Time Frame: Before surgery and up to 72 h reperfusion after surgery
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
Arbitrary units
  Before anesthesia | .07 (.04) | .11 (.04)
  After anesthesia | .06 (.04) | .12 (.04)
  10 min reperfusion | 1.22 (.08) | 1.37 (.08)
  20 min reperfusion | 1.14 (.09) | 1.3 (.09)
  3 h reperfusion | .52 (.08) | .53 (.08)
  6 h reperfusion | .21 (.04) | .22 (.04)
  24 h reperfusion | .05 (.03) | .09 (.01)
  72 h reperfusion | .03 (.01) | .03 (.01)

5. Secondary Outcome: Venous Plasma Cardiac Matrix Metalloproteinase-2 Activity Before and After Reperfusion
Description: Biochemical activity of MMP-2 activity in venous plasma, measured before surgery and up to 72h of reperfusion after surgery.
Time Frame: Before surgery and up to 72 h reperfusion after surgery
Measure: Mean (Standard Error); unit: Arbitrary units
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
Arbitrary units
  Before anesthesia | .99 (.05) | 1.06 (.05)
  After anesthesia | .93 (.04) | .96 (.04)
  10 min reperfusion | 1.01 (.06) | 1.05 (.06)
  20 min reperfusion | .87 (.04) | 1 (.04)
  3 h reperfusion | .99 (.05) | 1.06 (.05)
  6 h reperfusion | .92 (.07) | 1.07 (.07)
  24 h reperfusion | .78 (.05) | .9 (.05)
  72 h reperfusion | .78 (.04) | .9 (.04)

6. Secondary Outcome: Venous Plasma Concentration of Troponin-I
Description: Measurement of levels of TnI (troponin-I), a marker of cardiac cell damage
Time Frame: Before surgery and 10 minutes reperfusion after surgery
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
pg/ml
  Before surgery | 1.23 (.33) | 1.07 (.34)
  Post surgery | 1.39 (.46) | 1.78 (.47)

7. Secondary Outcome: Cleaved TroponinI/GAPDH Ratios in Right Atrial Biopsy
Description: Measurement of the ratios of cleaved TnI (troponin-I) versus GAPDH in biopsies collected from right atria. Measure is the ratio TnI/GAPDH
Time Frame: Before surgery and 10 minutes reperfusion after surgery
Measure: Mean (Standard Error); unit: Arbitrary units-Cleaved TnI/GAPDH
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
Arbitrary units-Cleaved TnI/GAPDH
  Before surgery | 1.1318 (.3852) | 2.3454 (.3978)
  Post surgery | 1.5195 (.3745) | 2.1893 (.3868)

8. Secondary Outcome: Venous Plasma Concentration of C-reactive Protein
Description: Measurement of inflammation marker C-reactive protein in plasma
Time Frame: Before surgery and up to 72 h reperfusion after surgery
Measure: Mean (Standard Error); unit: ng/ml
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
ng/ml
  Before anesthesia | 5.7 (2) | 10 (2)
  After anesthesia | 5.7 (1.8) | 9.9 (2)
  10 min reperfusion | 4 (1.3) | 7.5 (1.5)
  20 min reperfusion | 4 (1.5) | 7.2 (1.3)
  3 h reperfusion | 5.2 (1.7) | 9.4 (1.8)
  6 h reperfusion | 12.9 (2) | 16.3 (2.1)
  24 h reperfusion | 51 (1.9) | 48.8 (1.9)
  72 h reperfusion | 51.1 (1.2) | 51.2 (1.2)

9. Secondary Outcome: Venous Plasma Concentration of IL-6
Description: Measurement of inflammation marker interleukin-6 in plasma
Time Frame: Before surgery and up to 72 h reperfusion after surgery
Measure: Mean (Standard Error); unit: pg/ml
Arm/Group | Placebo Oral Tablet | Periostat
Number analyzed (Participants) | 22 | 20
pg/ml
  Before anesthesia | 5.7 (2) | 1.9 (2)
  After anesthesia | 5.6 (1.9) | 2.8 (1.9)
  10 min reperfusion | 15.4 (2.7) | 7.3 (2.7)
  20 min reperfusion | 24.4 (3.3) | 15.1 (3.4)
  3 h reperfusion | 72.9 (6.6) | 76.1 (6.7)
  6 h reperfusion | 75.6 (5.9) | 83.4 (6)
  24 h reperfusion | 66.4 (6.4) | 71.8 (6.5)
  72 h reperfusion | 39 (5.7) | 28.1 (5.8)

ADVERSE EVENTS:
Time Frame: 72 hours
Arm/Group | Placebo Oral Tablet | Periostat
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/20
Other Adverse Events (participants affected / at risk) | 0/22 | 0/20

LIMITATIONS AND CAVEATS:
Small sample size. LVSWI does not estimate diastolic dysfunction. Right atrial biopsies may not reflect changes in left ventricular MMP activity. Doxycycline dose- and time-response analyses is required to better assess the protective effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes